CLINICAL TRIAL: NCT06748703
Title: Optic Nerve Injury and the Effect of CPAP Treatment in Obstructive Sleep Apnea Patients
Brief Title: Optic Nerve Injury in Obstructive Sleep Apnea Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-204
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea (OSA); Ischemic Optic Neuropathy/Optic Nerve Stroke
Keywords: Obstructive Sleep Apnea; Nonarteritic Ischemic Optic Neuropathy; CPAP treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Optic Neuropathy, Ischemic | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP Treatment Group (Experimental): Patients with Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) who are eligible for CPAP therapy.
  Interventions: Device: CPAP Treatment

INTERVENTIONS:
Device: CPAP Treatment — CPAP therapy will be administered to patients for 3 months. The CPAP device will be set to deliver a continuous flow of air at a prescribed pressure to keep the patient's airway open during sleep.

SUMMARY:
Ischemic optic neuropathy (ION) is damage to the optic nerve caused by ischemia and hypoxia of the optic nerve due to an impairment of the blood supply to the optic nerve from the arteries. Obstructive Sleep Apnea Hypoventilation Syndrome (OSAHS) is a sleep-breathing disorder characterized by recurrent upper airway obstruction and apnea during sleep, leading to recurrent intermittent hypoxemia with fragmented sleep and daytime sleepiness. Due to the lack of accurate methods to evaluate blood flow, the correlation between the two is unclear and uncertain. The study will enroll 80 patients from the First Affiliated Hospital of Nanjing Medical University and categorize them into mild, moderate, and severe OSA groups according to their apnea-hypopnea index (AHI). Participants will undergo a baseline evaluation, including polysomnography (PSG) and ophthalmologic examinations such as optic nerve and macular blood flow OCT, visual acuity, refraction, intraocular pressure, and visual fields. Eligible patients will be treated with CPAP for 3 months, after which their PSG and ophthalmologic examination-related results will be re-evaluated to assess treatment efficacy.

DETAILED DESCRIPTION:
Ischemic optic neuropathy (ION) is damage to the optic nerve caused by ischemia and hypoxia in the optic nerve due to impairment of the blood supply of the arteries supplying the optic nerve. ION is an important blinding eye disease. It has been found that patients with OSAHS are often misdiagnosed as having normotensive glaucoma due to chronic hypoxia resulting in optic nerve ischemia and hypoxia, leading to the development of ION. However, the correlation between the two has been poorly studied and is uncertain due to the lack of accurate methods to evaluate blood flow.

The study will enroll 80 patients from the First Affiliated Hospital of Nanjing Medical University between the ages of 18-80 years. Participants will be diagnosed with OSA according to established guidelines and must be first-time visitors with no prior history of OSA surgery or CPAP treatment. Patients with severe cerebrovascular disease, psychiatric disorders, diagnosed diabetes mellitus with severe vascular complications, severe COPD, pulmonary hypertension, heart failure, or pregnancy will be excluded.

All participants will undergo a polysomnography (PSG) to determine the Apnea Hypopnea Index (AHI) and will be categorized into mild, moderate, or severe OSA groups. Ophthalmologic-related examinations will be performed to measure ocular parameters such as optic nerve and macular blood flow OCT, visual acuity, refraction, intraocular pressure (IOP), visual fields, and IOLMaster measurements of the eye axis.

Eligible patients will receive CPAP treatment for 3 months. After 3 months of CPAP treatment, participants will undergo another PSG examination with ophthalmologic correlation to re-evaluate sleep parameters and ocular parameters.

The collected data will be analyzed using SPSS software. Correlation analysis will be performed to assess the relationship between AHI, minimum SPO2, hypoxic load, respiratory load, blood pressure variability, heart rate variability, pulse wave amplitude decline index, ESS drowsiness score, and the following ophthalmologic parameters: optic nerve and macular blood flow OCT, visual acuity, refraction, intraocular pressure, visual field, and eye axis as measured by IOLMaster. Paired t-tests will be performed to analyze the changes in the above indexes before and after CPAP treatment; ANOVA with repeated measurements will be performed to analyze the long-term changes in the above indexes.

The aim of this study is to analyze the relationship between sleep apnea severity hypoxia indexes and ION in OSAHS patients. To analyze the improvement of ischemic optic neuropathy (ION) after 3 months of CPAP treatment and to establish a long-term cohort to observe the occurrence of ION in patients with OSA of different severities, as well as the improvement of ION with long-term CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 80 years.
2. Diagnosed with Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS)(apnea-hypopnea index≥5/h).
3. First-time diagnosis, with no previous surgical interventions or CPAP treatment for OSA.
4. Ability and willingness to provide informed consent for participation in the study.

Exclusion Criteria:

1. History of severe stroke or cerebral hemorrhage, or presence of neurological or psychiatric conditions that could affect study results.
2. Presence of active malignancies or other severe underlying diseases, such as severe liver or kidney dysfunction. Diagnosed with diabetes or other significant vascular diseases.
3. Presence of severe chronic obstructive pulmonary disease (COPD), severe asthma, severe pulmonary hypertension, or heart failure caused by any condition.
4. Pregnancy or having other conditions that make participation in this study unsuitable.
5. Extremely debilitated patients or those with severe underlying conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Optic nerve and macular blood flow | Baseline and 3 months of CPAP therapy
  Changes in optic nerve and macular blood flow in patients with OSA of varying severity were measured using blood flow optical coherence tomography (blood flow OCT).
Apnea Hypopnea Index (AHI) | Baseline and 3 months of CPAP therapy
  Number of apneas and hypoventilations per hour of sleep
Hypoxic Burden（HB） | Baseline and 3 months of CPAP therapy
  The sum of the area between the SpO2 trace and the desaturation baseline associated with all apnoea and hypopnoea events is divided by the total time of sleep.
Ventilatory burden | Baseline and 3 months of CPAP therapy
  The average ventilatory burden per event was defined as the multiplication of the average ventilation during the respiratory event and average duration of respiratory events. The total ventilatory burden for each participant was defined as the multiplication of respiratory event rate and average ventilatory area per event.
Blood pressure variability | Baseline and 3 months of CPAP therapy
  The main studies were on ultrashort-term variability (blood pressure variability between each heart beat) and short-term variability (blood pressure variability over a 24-hour period).
Heart rate variability | Baseline and 3 months of CPAP therapy
  Heart rate variability (HRV) is the variation of differences between consecutive cardiac cycles. For example, the standard deviation of NN intervals in 24 h (SDNN), the standard deviation of the mean of NN intervals per 5 min (SDANN), and the SDNN during wakefulness and sleep.
Pulse Wave Amplitude Drops Index | Baseline and 3 months of CPAP therapy
  The number of decreases (>30%) in pulse wave amplitude per hour detected by pulse oximetry based on photoplethysmographic volumetric tracing (PPG) signals during sleep.

SECONDARY OUTCOMES:
Time below 90% Saturation | Baseline and 3 months of CPAP therapy
  Percentage of total time with oxygen saturation below 90% of total monitoring time.
Lowest SpO2 at night | Baseline and 3 months of CPAP therapy
  The lowest SpO2 value recorded during the nightly test.
Mean SpO2 | Baseline and 3 months of CPAP therapy
  Mean SpO2 values during nighttime monitoring.
Oxygen Desaturation Index | Baseline and 3 months of CPAP therapy
  The number of oxygen desaturation events per hour of sleep.The desaturation thresholds of 3% (ODI3) or 4% (ODI4) are commonly chosen in the analysis of OSA.
Vision | Baseline and 3 months of CPAP therapy
  The patient's naked eye visual acuity in the right and left eyes was checked using a visual acuity chart.
Diopter | Baseline and 3 months of CPAP therapy
  Qualitative and quantitative analysis of the refractive status of the eye under test using computerized optometry.
Intraocular pressure | Baseline and 3 months of CPAP therapy
  Measurement of intraocular pressure (IOP) in the eye under test using a non-contact tonometer.
Field of view | Baseline and 3 months of CPAP therapy
  An automated visual field meter was used to detect the total loss of the visual field and the extent and depth of limiting defects in the tested eye.
Axon of the eye | Baseline and 3 months of CPAP therapy
  The IOLMaster was utilized to measure the eye axis of the tested eye.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. The informed consent will be ansigned before enrolled in the study and ensured to keep personal information confidential.